CLINICAL TRIAL: NCT05542693
Title: Phase IIb, Randomized, Double-blind, Non-inferior, Multicenter Study to Evaluate the Safety and Immunogenicity of the Self-replicating Nanoparticle Carrier Replicon RNA Carrier (repRNA) Vaccine in Adults 18 to 65 Years of Age
Brief Title: Safety and Immunogenicity of the RNA MCTI CIMATEC HDT Vaccine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azidus Brasil (Industry)
Collaborators: SENAI CIMATEC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RNA-MCTI-CIMATEC-HDT-002
Record Dates: First submitted 2022-08-26; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: COVID-19; COVID-19 Vaccine
MeSH Terms: conditions — COVID-19 | interventions — repRNA-CoV2S vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RNA MCTI CIMATEC HDT 5µg (Experimental): Intramuscular injections of novel Lipid-Inorganic Nanoparticle (LION) formulated replicating RNA-based vaccine (VACCINE RNA MCTI CIMATEC HDT) at a dose of 5 µg of single-dose administration on day 1.
  Interventions: Biological: RNA MCTI CIMATEC HDT 5µg
- RNA MCTI CIMATEC HDT 10µg (Experimental): Intramuscular injections of novel Lipid-Inorganic Nanoparticle (LION) formulated replicating RNA-based vaccine (VACCINE RNA MCTI CIMATEC HDT) at a dose of 10 µg of single-dose administration on day 1.
  Interventions: Biological: RNA MCTI CIMATEC HDT 10µg
- Covishield® - AstraZeneca (Active Comparator): Intramuscular injections of vaccine Covishield® - AstraZeneca at a usual dose of single-dose administration on day 1.
  Interventions: Biological: Covishield® - AstraZeneca
- Comirnaty® - Pfizer (Active Comparator): Intramuscular injections of vaccine Comirnaty® - Pfizer at a usual dose of single-dose administration on day 1.
  Interventions: Biological: Comirnaty® - Pfizer

INTERVENTIONS:
Biological: RNA MCTI CIMATEC HDT 5µg — Adults previously immunized will be randomized to receive a single booster vaccine: experimental (MCTI-CIMATEC-HDT RNA)
  Arms: RNA MCTI CIMATEC HDT 5µg
Biological: RNA MCTI CIMATEC HDT 10µg — Adults previously immunized will be randomized to receive a single booster vaccine: experimental (MCTI-CIMATEC-HDT RNA)
  Arms: RNA MCTI CIMATEC HDT 10µg
Biological: Covishield® - AstraZeneca — Adults previously immunized will be randomized to receive a single booster vaccine comparator (Comirnaty - Pfizer)
  Arms: Covishield® - AstraZeneca
Biological: Comirnaty® - Pfizer — Adults previously immunized will be randomized to receive a single booster vaccine comparator (Comirnaty - Pfizer and (Covishield - Oxford/Astrazen).
  Arms: Comirnaty® - Pfizer

SUMMARY:
A multicenter, randomized, double-blind, active comparator, non-inferiority, multicenter IIb clinical trial to compare the safety and immunogenicity of two dose levels of the MCTI CIMATEC HDT RNA Vaccine against two authorized COVID-19 vaccines in Brazil (Comirnaty - Pfizer and Covishield - Oxford/AstraZeneca) in 300 participants. Each vaccine will be provided as a single booster vaccine in adults aged 18 to 65 years previously immunized with both vaccines (Comirnaty - Pfizer and Covishield - Oxford/Astrazen). The investigational product MCTI C HDT will be administered in one of the two doses evaluated (5µg and 10 µg). The comparator products will be Comirnaty - Pfizer and Covishield - Oxford/AstraZeneca. The primary outcomes will be the number of participants with a 2-fold increase or more on average by titers of neutralizing D64G pseudovirus strain (pNT50) and comparison of titers generated by 5µg and 10µg doses of MCTI-CIMATEC-HDT RNA Vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Complete primary vaccination with Cominarty (Pfizer) or Covishield (Oxford/Astrazeneca) vaccines, and at least one booster dose with Cominarty (Pfizer) or Covishield (Oxford/Astrazeneca) vaccines. The last duration being at least 4 before the study duration.
3. Adult in a healthy condition or with a stable health status if pre-existing medical history.
4. Sign informed consent, be able and willing to make the assessment, be accessible by telephone or in person by the local study team and willing to remain in the study area for the duration of the study
5. For women of childbearing age: a highly negative sensitive urinary pregnancy test during the inclusion visit AND use an effective contraceptive method.

Exclusion Criteria:

1. History of COVID-19 in the 30 days before study enrollment.
2. Participation in other clinical studies in the last 12 (two) months.
3. Receive or plan any immunization during the study, except the seasonal influenza vaccine, within 30 days of enrollment.
4. Receive a blood or immunoglobulin transfusion within 90 days before study enrollment;
5. Blood donation up to 30 days before inclusion in the study;
6. Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immunomodulatory drugs.
7. History of autoimmune disease or immunosuppression.
8. Rash, tattoos, or any other skin condition that could adversely affect the vaccine injection site.
9. Body mass index (BMI) > 35.
10. Known or suspected drug or alcohol abuse in the last 6 months;
11. History of previous anaphylaxis or severe allergic reactions to the vaccine, products known to contain polyethene glycol (PEG) or unknown allergens.
12. History of myocarditis or carditis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity of the RNA MCTI CIMATEC HDT Vaccine (Non-inferiority) | Day 29 after vaccination until day 181.
  Proportion of participants with a 2-fold or greater increase in geometric mean neutralizing antibody titers against D614G pseudovirus strain (pNT50).
Immunogenicity of the RNA MCTI CIMATEC HDT Vaccine (Dose determination) | Day 29 after vaccination until day 181.
  Comparison of antibody titers generated by 5µg and 10µg doses of the MCTI-CIMATEC-HDT RNA Vaccine

IPD SHARING:
Plan to Share IPD: No